CLINICAL TRIAL: NCT03406195
Title: Modulation of Episodic Memory Using Theta Burst Stimulation (TBS)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants recruited, IRB closed
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00086794
Record Dates: First submitted 2018-01-16; First posted 2018-01-23 (Actual); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Aging
Keywords: transcranial magnetic stimulation
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: We will perform episodic memory task before and after the TMS session
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- healthy older adults (Experimental): Healthy older adults who will receive TMS
  Interventions: Device: Transcranial magnetic stimulation (TMS)

INTERVENTIONS:
Device: Transcranial magnetic stimulation (TMS) — TMS paradigm called theta burst stimulation

SUMMARY:
The goal of this study is to evaluate the effect of white matter guided theta burst stimulation on episodic memory task performance in healthy older adults. The investigators aim to propagate the effect of theta burst stimulation from a superficial locus of stimulation (angular gyrus) to hippocampus and parahippocampal regions using white matter tract connection between these regions. Study activities and population group - for the study plans to recruit 20 healthy older adults who already have white matter scans acquired as part of another study performed by the Cabeza Lab at Duke University.

Using tractography the exact site of stimulation on the cortical surface will be localized. An initial motor evoked potential (MEP) assessment will differentiate responders to theta burst stimulation from non responders. Responders will receive 1200 pulses of intermittent theta burst stimulation (iTBS) or sham stimulation to the angular gyrus while they perform the encoding portion of an episodic memory task. There after, they will perform retrieval piece of the task and data analysis will compare these performances.

DETAILED DESCRIPTION:
Aims and Hypotheses The purpose of the study is to evaluate the effect of theta burst stimulation (TBS) which is a relatively new paradigm of transcranial magnetic stimulation (TMS) on episodic memory (EM) in healthy older adults (hOA).

Aim1: Evaluate the effect of theta burst stimulation (TBS) on episodic memory (EM) in healthy older adults. Hypothesis 1 - There will be significant improvement in EM compared to baseline with one session of TBS.

Aim 2: Correlate white matter integrity to improvement in task retrieval with TBS. Hypothesis 2- Stronger white matter (WM) tract connections correlate to greater improvement in retrieval performance.

BACKGROUND Alzheimer's disease (AD) affects 5 million Americans, at a cost of over 200 billion dollars. The first and most debilitating symptom of AD is a severe deficit in the ability to remembering personal past events, or episodic memory (EM), which eventually renders patients isolated from family and friends and unable to live independently. This EM deficit reflects primarily the deterioration of medial temporal lobe regions, particularly the hippocampus (HC). AD treatments must start very early in the disease progression, when brain damage is still small, and the earliest stage when AD can be diagnosed is known as mild cognitive impairment due to AD (MCI-AD).

Recently, different forms of noninvasive brain stimulation techniques have been applied to healthy older adults, AD and MCI-AD to improve memory impairment. Most of these trials used high-frequency repetitive transcranial magnetic stimulation (rTMS) applied to the left dorsolateral prefrontal cortex (DLPFC). Although a small number of these studies have shown beneficial effects, considerable questions remain as to whether TMS has clinically relevant effects in elderly populations, as well as to what neuroscience-based mechanisms account for these effects. An obstacle for using TMS to enhance EM is that the brain region most critical for EM and most affected by early AD, the hippocampus (HC), is situated deep inside the brain, beyond TMS direct effects (~1" below the skull). One study attempted to target hippocampus and peri-hippocampal regions for stimulation via TMS. They stimulated the lateral parietal cortex and utilized functional connectivity between this region and hippocampus/peri-hippocampal regions (mainly entorhinal cortex) to enhance performance on an associative memory task. The inferior longitudinal fasciculus connects angular gyrus to hippocampus and para-hippocampal regions, and could propagate stimulation effects from cortical to subcortical structures, although studies on effect on TMS on white matter neuronal populations are limited as detailed below. The effect of TMS on neuronal populations in the white matter tracts was recently modeled using tractography and e-field calculations, and increasingly, these approaches need to account for what percentage of variance in motor threshold (MT) would be accounted for by white matter tracts.

TBS is a potent paradigm of TMS. As detailed in a seminal paper by Huang et al, there are 2 patterns for the paradigm: - continuous theta burst stimulation (cTBS) and intermittent theta burst stimulation (iTBS). The former produces suppression of MEP and the latter produces increase in MEP. iTBS delivers 50 Hz stimuli in packets of 10 lasting 2 seconds. Each stimulus burst delivered at 50 Hz is given every 200 milliseconds making the overall frequency of stimulus delivery 5 Hz. Hence the stimulation encompasses nested 50 Hz bursts (gamma frequency) given at 5 Hz (theta frequency). Most investigational studies which did not have treatment outcome measures have used either 40 second of cTBS or 190 seconds of iTBS. Both these paradigms have been shown to cause changes in MEP for 60 minutes. Variations in pattern of stimulation have also been effective, although there are limited studies to warrant its use. The investigators therefore propose to use stimulate the function of the hippocampal formation in healthy older adults (hOA) by targeting a cortical region directly connected to the hippocampal formation: the angular gyrus. To increase indirect effects on hippocampal formation, the investigators will use the most powerful TMS technique available, intermittent Theta Burst Stimulation (iTBS).

METHODOLOGY The study is designed to be a pilot one evaluating the effect of TBS on EM in healthy older adults (hOA). The investigators plan to screen 30 participants to select 20 subjects.

Screening Potential participants will be in the age group of 60-80 years and encompasses subjects who have been recruited to previous studies at Cabeza Lab (Pro00005021), hence having brain imaging data already collected.

Study procedure On day 1 of the study, subjects will have the National Institute of Health (NIH) Toolbox administered to them. The NIH toolbox is a comprehensive set of neuro-behavioral measurements that quickly assesses cognitive functions from the convenience of an iPad. Total time allotted for NIH toolbox administration is 45 minutes. Following this, subjects will have motor evoked potential (MEP) performed after which they will be administered intermittent theta burst stimulation (iTBS) to motor cortex. This will be followed by measurement of motor evoked potential (MEP) again. Subjects who do not show a 10 % increase in motor evoked potential (MEP) with iTBS will be excluded from further parts of the study.

Our study uses a specific kind of TMS, known as intermittent theta burst stimulation (iTBS). On day 1 of the study, subjects will be administered either left-sided iTBS to the motor cortex. The subject will be seated in a chair. Electromyogram (EMG) electrodes will be applied to the right hand for motor evoked potential (MEP) recording. For iTBS the active motor threshold would be 80 % as used in most theta burst studies detailed in this review. Subjects would receive iTBS comprising 50 Hz bursts given at 3 to 5 Hz for close to 3 minutes which comprises 19 trains and 600 pulses. The subject will be monitored until MEPs return to baseline. A side effects checklist will be completed at the beginning and at the end of the experimental session. All sessions will be performed by one of the protocol investigators, or by a trained and accredited research assistant supervised by the protocol investigators.

If a 10 % increase is seen in the MEP, then subjects will receive a second session of iTBS or sham stimulation to the left angular gyrus one hour after the screening session. If they receive iTBS, this will comprise 6 minutes of stimulation equivalent to 1200 pulses and 38 trains of the stimulus. The subject will be monitored until MEPs return to baseline. A side effects checklist will be completed at the beginning and at the end of the experimental session. Sham stimulation will use superficial electrodes to mimic the experience of receiving actual stimulation. All sessions will be performed by one of the protocol investigators, or by a trained and accredited research assistant supervised by the protocol investigators. Subjects will perform encoding trials of episodic memory task with stimulation and retrieval piece of the task after the stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy controls in the age group 60-80 years old
* No other Diagnostic and Statistical Manual of Mental Disorders (DSM) 5 axis 1 diagnoses
* Willing to provide informed consent
* Structural magnetic resonance imaging (MRI) and diffusion tensor imaging (DTI) data available

Exclusion Criteria:

* Subjects are unable or unwilling to give informed consent
* Presence of any organic brain illness
* Presence or history of stroke, traumatic brain injury or head injury with loss of consciousness, transient ischemic attack (TIA), any diagnosed neurological disorder including but not limited to multiple sclerosis, Huntington's disease, Parkinson's disease, dementia or major neurocognitive disorder.
* Presence of cranial metal implants, structural brain lesion including but not limited to cerebral aneurysms.
* Presence of devices that may be affected by repetitive transcranial magnetic stimulation (rTMS) (pacemaker, medication pump, cochlear implant, implanted brain stimulator)
* Current or recent (within the past 6 months) substance abuse or dependence, excluding nicotine and caffeine.
* Current serious medical illness
* History of seizure except those therapeutically induced by electroconvulsive therapy (ECT) (childhood febrile seizures are acceptable and these subjects may be included in the study), history of epilepsy in self or first degree relatives
* For subjects age > 59 years, a total scaled score < 8 on the Dementia Rating Scale-2.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-12-15 (Estimated); Primary Completion 2019-12-30 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
Episodic memory retrieval task decision | 40 minutes
  Four-choice decision (1- definitely there is a link, 2-probably there is a link, 3-probably there is no link, 4-definitely there is no link) in response to semantic link retrieval between 2 words

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Cabeza, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Trebbastoni A, Pichiorri F, D'Antonio F, Campanelli A, Onesti E, Ceccanti M, de Lena C, Inghilleri M. Altered Cortical Synaptic Plasticity in Response to 5-Hz Repetitive Transcranial Magnetic Stimulation as a New Electrophysiological Finding in Amnestic Mild Cognitive Impairment Converting to Alzheimer's Disease: Results from a 4-year Prospective Cohort Study. Front Aging Neurosci. 2016 Jan 12;7:253. doi: 10.3389/fnagi.2015.00253. eCollection 2015. PMID 26793103
- [Background] Julkunen P, Jauhiainen AM, Westeren-Punnonen S, Pirinen E, Soininen H, Kononen M, Paakkonen A, Maatta S, Karhu J. Navigated TMS combined with EEG in mild cognitive impairment and Alzheimer's disease: a pilot study. J Neurosci Methods. 2008 Jul 30;172(2):270-6. doi: 10.1016/j.jneumeth.2008.04.021. Epub 2008 Apr 29. PMID 18533272
- [Background] Elder GJ, Taylor JP. Transcranial magnetic stimulation and transcranial direct current stimulation: treatments for cognitive and neuropsychiatric symptoms in the neurodegenerative dementias? Alzheimers Res Ther. 2014 Nov 10;6(9):74. doi: 10.1186/s13195-014-0074-1. eCollection 2014. PMID 25478032
- [Background] Drumond Marra HL, Myczkowski ML, Maia Memoria C, Arnaut D, Leite Ribeiro P, Sardinha Mansur CG, Lancelote Alberto R, Boura Bellini B, Alves Fernandes da Silva A, Tortella G, Ciampi de Andrade D, Teixeira MJ, Forlenza OV, Marcolin MA. Transcranial Magnetic Stimulation to Address Mild Cognitive Impairment in the Elderly: A Randomized Controlled Study. Behav Neurol. 2015;2015:287843. doi: 10.1155/2015/287843. Epub 2015 Jun 16. PMID 26160997
- [Background] Wang JX, Rogers LM, Gross EZ, Ryals AJ, Dokucu ME, Brandstatt KL, Hermiller MS, Voss JL. Targeted enhancement of cortical-hippocampal brain networks and associative memory. Science. 2014 Aug 29;345(6200):1054-7. doi: 10.1126/science.1252900. PMID 25170153
- [Background] Rushworth MF, Behrens TE, Johansen-Berg H. Connection patterns distinguish 3 regions of human parietal cortex. Cereb Cortex. 2006 Oct;16(10):1418-30. doi: 10.1093/cercor/bhj079. Epub 2005 Nov 23. PMID 16306320
- [Background] Uddin LQ, Supekar K, Amin H, Rykhlevskaia E, Nguyen DA, Greicius MD, Menon V. Dissociable connectivity within human angular gyrus and intraparietal sulcus: evidence from functional and structural connectivity. Cereb Cortex. 2010 Nov;20(11):2636-46. doi: 10.1093/cercor/bhq011. Epub 2010 Feb 12. PMID 20154013
- [Background] Huang YZ, Edwards MJ, Rounis E, Bhatia KP, Rothwell JC. Theta burst stimulation of the human motor cortex. Neuron. 2005 Jan 20;45(2):201-6. doi: 10.1016/j.neuron.2004.12.033. PMID 15664172
- [Background] Wischnewski M, Schutter DJ. Efficacy and Time Course of Theta Burst Stimulation in Healthy Humans. Brain Stimul. 2015 Jul-Aug;8(4):685-92. doi: 10.1016/j.brs.2015.03.004. Epub 2015 Mar 26. PMID 26014214
- [Background] Suppa A, Huang YZ, Funke K, Ridding MC, Cheeran B, Di Lazzaro V, Ziemann U, Rothwell JC. Ten Years of Theta Burst Stimulation in Humans: Established Knowledge, Unknowns and Prospects. Brain Stimul. 2016 May-Jun;9(3):323-335. doi: 10.1016/j.brs.2016.01.006. Epub 2016 Jan 27. PMID 26947241
- [Background] Davis SW, Dennis NA, Buchler NG, White LE, Madden DJ, Cabeza R. Assessing the effects of age on long white matter tracts using diffusion tensor tractography. Neuroimage. 2009 Jun;46(2):530-41. doi: 10.1016/j.neuroimage.2009.01.068. PMID 19385018
- [Background] Davis SW, Kragel JE, Madden DJ, Cabeza R. The architecture of cross-hemispheric communication in the aging brain: linking behavior to functional and structural connectivity. Cereb Cortex. 2012 Jan;22(1):232-42. doi: 10.1093/cercor/bhr123. Epub 2011 Jun 7. PMID 21653286
- [Background] Kier EL, Staib LH, Davis LM, Bronen RA. MR imaging of the temporal stem: anatomic dissection tractography of the uncinate fasciculus, inferior occipitofrontal fasciculus, and Meyer's loop of the optic radiation. AJNR Am J Neuroradiol. 2004 May;25(5):677-91. PMID 15140705
- [Background] Kier EL, Staib LH, Davis LM, Bronen RA. Anatomic dissection tractography: a new method for precise MR localization of white matter tracts. AJNR Am J Neuroradiol. 2004 May;25(5):670-6. PMID 15140704
- [Background] Oberman L, Edwards D, Eldaief M, Pascual-Leone A. Safety of theta burst transcranial magnetic stimulation: a systematic review of the literature. J Clin Neurophysiol. 2011 Feb;28(1):67-74. doi: 10.1097/WNP.0b013e318205135f. PMID 21221011
- [Background] Daselaar SM, Fleck MS, Dobbins IG, Madden DJ, Cabeza R. Effects of healthy aging on hippocampal and rhinal memory functions: an event-related fMRI study. Cereb Cortex. 2006 Dec;16(12):1771-82. doi: 10.1093/cercor/bhj112. Epub 2006 Jan 18. PMID 16421332
- [Background] Rossi S, Hallett M, Rossini PM, Pascual-Leone A; Safety of TMS Consensus Group. Safety, ethical considerations, and application guidelines for the use of transcranial magnetic stimulation in clinical practice and research. Clin Neurophysiol. 2009 Dec;120(12):2008-2039. doi: 10.1016/j.clinph.2009.08.016. Epub 2009 Oct 14. PMID 19833552
- [Background] Wassermann EM. Risk and safety of repetitive transcranial magnetic stimulation: report and suggested guidelines from the International Workshop on the Safety of Repetitive Transcranial Magnetic Stimulation, June 5-7, 1996. Electroencephalogr Clin Neurophysiol. 1998 Jan;108(1):1-16. doi: 10.1016/s0168-5597(97)00096-8. PMID 9474057
- [Background] Loo C, Sachdev P, Elsayed H, McDarmont B, Mitchell P, Wilkinson M, Parker G, Gandevia S. Effects of a 2- to 4-week course of repetitive transcranial magnetic stimulation (rTMS) on neuropsychologic functioning, electroencephalogram, and auditory threshold in depressed patients. Biol Psychiatry. 2001 Apr 1;49(7):615-23. doi: 10.1016/s0006-3223(00)00996-3. PMID 11297719